CLINICAL TRIAL: NCT00525122
Title: Treatment of M.Graves With Radioactive Iodine: Follow-up Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medisch Centrum Rijnmond-Zuid, Netherlands (Other Government)
Responsible Party: A. Berghout, MCRZ
Other Study IDs: 2006/60
Record Dates: First submitted 2007-09-04; First posted 2007-09-05 (Estimated); Last update posted 2008-05-22 (Estimated); Status verified 2008-05

CONDITIONS: Hyperthyroidism
Keywords: hyperthyroidism; radioactive iodine; antithyroid drugs; Hyperthyroidism, treatment with radioactive iodine without antithyroid drugs
MeSH Terms: conditions — Hyperthyroidism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients with hyperthyroidism who are will be treated with radioactive iodine.

SUMMARY:
Hypothesis: What is the natural course after treatment with radioactive iodine in patients with hyperthyroidism?

What are the determinants for the development of acute hypo- or hyperthyroidism after treatment with radioactive iodine without antithyroid drugs?

ELIGIBILITY:
Inclusion Criteria:

* Patients wth hyperthyroidism who are eligible for treatment with radioactive iodine
* Age > 18 years

Exclusion Criteria:

* Severe ophthalmopathy
* Pregnancy or wish to pregnancy on short term
* Breastfeeding
* Patients already treated with radioactive iodine
* Known cardiovascular diseases or other severe comorbidity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of 18 years and older with hyperthyroidism who are eligible for treatment with radioactive iodine.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2007-09

CONTACTS AND LOCATIONS:
Overall Officials: A. Berghout, MD, PhD, Principal Investigator — Medisch Centrum Rijnmond-Zuid, Netherlands; C. van Noord, MD, Principal Investigator — Medisch Centrum Rijnmond-Zuid, Netherlands
Locations (1):
- MCRZ, Rotterdam, South Holland, Netherlands